CLINICAL TRIAL: NCT01407497
Title: A Phase I Trial to Assess Safety and Immunogenicity of i.d. DNA Priming and i.m. MVA Boosting in Healthy Volunteers in Mozambique and to Develop Further HIV Vaccine Trial Capacity Building in Mozambique
Brief Title: Safety and Immunogenicity Study of a DNA Priming and MVA Boosting Strategy of HIV Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Instituto Nacional de Saúde, Mozambique (Other Government)
Collaborators: Swedish Institute for Communicable Disease Control, Sweden (Unknown); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TAMOVAC-01-MZ
Record Dates: First submitted 2011-08-01; First posted 2011-08-02 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: HIV Infections
Keywords: HIV; Vaccine; DNA; Prevention
MeSH Terms: conditions — HIV Infections | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IA (Active Comparator): 600 µg i.d. (separate plasmids pools) of DNA priming at weeks 0, 4 and 12 108 pfu i.m. MVA boosting at weeks 24 and 36
  Interventions: Biological: DNA HIVIS and MVA-CMDR
- IB (Placebo Comparator): 2 x 0.1 ml of saline solution i.d at weeks 0, 4 and 12 saline solution i.m at weeks 24 and 36
  Interventions: Biological: Saline solution
- IIA (Active Comparator): 1200 µg i.d. (separate plasmids pools) of DNA priming at weeks 0, 4 and 12;108 pfu i.m. MVA boosting at weeks 24 and 36
  Interventions: Biological: DNA HIVIS and MVA-CMDR
- IIB (Placebo Comparator): 2 x 0.2 ml of saline solution i.d at weeks 0, 4 and 12 ; saline solution i.m at weeks 24 and 36
  Interventions: Biological: Saline solution

INTERVENTIONS:
Biological: DNA HIVIS and MVA-CMDR — 600 µg i.d. (separate plasmids pools) of DNA priming at weeks 0, 4 and 12; 108 pfu i.m. MVA boosting at weeks 24 and 36
  Arms: IA
Biological: DNA HIVIS and MVA-CMDR — 1200 µg i.d. (separate plasmids pools) of DNA priming at weeks 0, 4 and 12 ; 108 pfu i.m. MVA boosting at weeks 24 and 36
  Arms: IIA
Biological: Saline solution — 2 x 0.1 ml of saline solution i.d at weeks 0, 4 and 12 ; saline solution i.m at weeks 24 and 36
  Arms: IB
Biological: Saline solution — 2 x 0.2 ml of saline solution i.d at weeks 0, 4 and 12 ; saline solution i.m at weeks 24 and 36
  Arms: IIB

SUMMARY:
While antiretroviral drugs have shown great promise in reducing HIV replication and thus in reducing HIV/AIDS associated morbi-mortality and HIV transmission, the cost is substantial and side effects are a potentially limiting factor. Development of an effective safe-affordable vaccine is likely to be the best way to stop further virus spread. The study aims to determine safety and immunogenicity of the DNA-vaccine at a dose of 600µg and 1200µg delivered id in combination with MVA-CMDR boost im.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 26 years
2. Willing to undergo HIV (Human Immunodeficiency Virus) counseling and testing
3. Have a negative antigen/antibody or antibody ELISA for HIV infection
4. Able to give informed consent
5. Satisfactory completion of an assessment of understanding prior to enrolment defined as 89% correct answers after three opportunities to take the test
6. Basic abilities to read and write
7. Resident in Maputo, and willing to remain so for the duration of the study
8. At low risk of HIV infection, defined as the absence of an identifiable risk factor/ behavior (their presence is therefore an exclusion criteria):

   * sexual partner with HIV
   * sexual partner with unknown HIV serostatus who is also unwilling to use protective condoms consistently in all sexual relations
   * sexual partner is known to be at high risk for HIV
   * more than one sexual partner in the last 6 months
   * history of being an alcoholic [as medically defined or more than 35 units /week]
   * history of Sexually Transmitted Infection (STI) within past 6 months
9. Verbal assurances that adequate birth control methods are used not to conceive/father a child during the study and up to 3 months after the last vaccine injection.
10. Women shall have a negative urine pregnancy test
11. Be willing to practice safe sex for the duration of the study to avoid sexually transmitted infections including HIV
12. Good health as determined by medical history, physical examination, clinical judgment and by key laboratory parameters as judged by the study physician.
13. Laboratory criteria:

    * Hemoglobin >10.5g/dl
    * White blood cell count <13,000/mm3
    * Neutrophils >1,300/mm3
    * Lymphocytes >1.000/ mm3
    * Platelets >120,000/ mm3
    * Random Blood Glucose < 6.44 mmol/L; if elevated, then a Fasting Blood Glucose < 6.11mmol/L (according to DAIDS Table for Lab Criteria)
    * Bilirubin <1.25 x uln
    * Alanine transaminase (ALT) <1.25 x uln
    * Urine dipstick for protein and blood: negative or trace. (If either is ¿ 1+, complete urinalysis (UA) will be performed.

Exclusion Criteria:

1. At risk of HIV infection as mentioned above in the inclusion criteria
2. Active tuberculosis or other systemic infectious process elicited by review of systems, physical examination and laboratory detection
3. A history of immunodeficiency, chronic illness requiring continuous or frequent medical intervention
4. Autoimmune disease by history and physical examination
5. Hives or recurrent hives and severe eczema
6. A history of psychiatric, medical (including traditional medicine) and/or substance abuse problems during the past 6 months that the investigator believes would adversely affect the volunteer's ability to participate in the trial
7. History of epilepsy, or currently taking anti-epileptics
8. Received blood or blood products or immunoglobulins in the past 3 months
9. Receiving immunosuppressive therapy such as systemic corticosteroids or cancer chemotherapy
10. Use of experimental therapeutic agents within 30 days of study entry
11. Reception of any live, attenuated vaccine within 60 days of study entry.
12. Abnormality in Electrocardiogram (ECG) that could indicate risk or make interpretation of vaccine effects difficult according to the study operating procedures
13. Previously received an HIV vaccine candidate
14. History of severe local or general reaction to vaccination defined as:

    * Local: Extensive, indurate redness and swelling involving most of the major circumference of the arm, not resolving within 72 hours
    * General: Fever >= 39.5 0C within 48 hours; anaphylaxis; bronchospasm; laryngeal edema; collapse; convulsions or encephalopathy within 72 hours
15. Being a lactating mother
16. Study site employees who are involved in the protocol and may have direct access to the immunogenicity results
17. Unlikely to comply with protocol as judged by the principal investigator or his designate.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-08; Primary Completion 2013-03 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Adverse events (local and system reactogenicity) | 44 weeks
  The safety of immunization will be assessed by clinical features and standard clinical chemistry and hematological tests. Safety endpoints: Adverse events will be assessed using a standard format for soliciting local and systemic reactogenicity to the vaccine and collection of unsolicited adverse events. Solicited reactogenicity will be evaluated for 7 days following each vaccination. All other AE will be collected from the time of first injection until the end of the study follow-up period.
Immunogenicity | 44 weeks
  The primary immunogenicity endpoint will be determined by the interferon gamma (IFN-gama) enzyme linked immunospot (ELISPOT) assay.
  Secondary immunogenicity endpoints will include cellular immune responses determined by intracellular cytokine staining and T cell proliferation assays as well as binding antibody and neutralizing antibody responses.

CONTACTS AND LOCATIONS:
Overall Officials: Ilesh Jani, PhD, Principal Investigator — Instituto Nacional de Saúde, Mozambique; Nafissa Osman, MD, PhD, Principal Investigator — Hospital Central de Maputo
Locations (1):
- Centro de Investigação e Treino em Saúde de Polana Caniço, Maputo, Cidade de Maputo, Mozambique

REFERENCES:
- [Derived] Viegas EO, Tembe N, Nilsson C, Meggi B, Maueia C, Augusto O, Stout R, Scarlatti G, Ferrari G, Earl PL, Wahren B, Andersson S, Robb ML, Osman N, Biberfeld G, Jani I, Sandstrom E. Intradermal HIV-1 DNA Immunization Using Needle-Free Zetajet Injection Followed by HIV-Modified Vaccinia Virus Ankara Vaccination Is Safe and Immunogenic in Mozambican Young Adults: A Phase I Randomized Controlled Trial. AIDS Res Hum Retroviruses. 2018 Feb;34(2):193-205. doi: 10.1089/AID.2017.0121. Epub 2017 Nov 27. PMID 28969431